CLINICAL TRIAL: NCT06224855
Title: An Open-label Dose Escalation and Cohort Expansion Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and and Efficacy of DXC006 in Patients With Advanced Solid Tumors and Hematologic Malignancies
Brief Title: A Study of DXC006 in Patients With Advanced Solid Tumors and Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou DAC Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DXC006-001
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumors; Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose 1:Drug(DXC006), Dose 2:Drug(DXC006), Dose 3:Drug(DXC006), Dose 4:Drug(DXC006), Dose 5:Drug(DXC006), Dose 6:Drug(DXC006).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Dose Escalation DXC006, Cohort Expansion DXC006
  Interventions: Drug: DXC006

INTERVENTIONS:
Drug: DXC006 — Dose escalation period: DXC006 is administered intravenously every two weeks (Q2W) at the dose corresponding to the enrolled dose cohort.
  Dose expansion period: DXC006 is administered intravenously Q2W at the corresponding dose.
  Other Names: Recombinant Humanized Antibody-drug conjugate

SUMMARY:
This is a phase I, open-label, first-in-human clinical study designed to evaluate the safety, tolerability, MTD, DLT, RP2D, the PK characteristics, preliminary anti-tumor activity, the immunogenicity of DXC006 in patients with a variety of solid tumors, including small cell lung cancer, multiple myeloma, and neuroblastoma, and hematological malignancies.

DETAILED DESCRIPTION:
This is a phase I, open-label, first-in-human clinical study designed to evaluate the safety, tolerability, MTD, DLT, RP2D, the PK characteristics, preliminary anti-tumor activity, the immunogenicity of DXC006 in patients with a variety of solid tumors, including small cell lung cancer, multiple myeloma, and neuroblastoma, and hematological. malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily signed the informed consent form and followed the protocol requirements.
2. Gender is not limited.
3. Age ≥ 18 years old.
4. Expected survival time ≥ 3 months.
5. The Eastern Cooperative Oncology Group (ECOG) score 0-2.
6. Subjects may provide biopsy or archival tumor tissue samples for the central laboratory to confirm expression levels of Target protein.
7. Patients with solid tumors or hematologic tumors who have failed standard therapy, including small cell lung cancer, multiple myeloma, neuroblastoma, etc..
8. Patients who have received ASCT treatment must meet the following conditions:

   1. ASCT > 100 days from start of study treatment.
   2. no active infection.
9. Toxicity from prior antineoplastic therapy has recovered to Grade ≤ 1 (except alopecia) as defined by NCI-CTCAE v5.0, including peripheral neuropathy ≤ Grade 2.
10. Organ function must meet the following requirements: blood routine:

(1) Patients with multiple myeloma: absolute neutrophil count (ANC) ≥ 1.0×109/L (previous use of granulocyte colony-stimulating factor [G-CSF] is allowed, and G-CSF is not allowed within 7 days before laboratory examination during the screening period);Platelet count ≥ 50×109/L (platelet transfusion is not allowed within 7 days before laboratory tests during the screening period).

Hemoglobin (HGB) ≥ 75 g/L (prior red blood cell [RBC] transfusions or recombinant human erythropoietin are allowed; Within 7 days before the laboratory examination during the screening period, red blood cell transfusion is not allowed).

(2) Other patients: Absolute neutrophil count (ANC) ≥ 1.5×109/L, Platelet count ≥ 100×109/L, Hemoglobin (HGB) ≥ 90 g/L Liver: total bilirubin (TBIL) ≤ 1.5×ULN, except for subjects with congenital bilirubinemia, such as Gilbert's syndrome (direct bilirubin ≤ 1.5×ULN); Glutamate aminotransferase (AST) and alanine aminotransferase (ALT) both ≤ 3.0×ULN.

In the presence of liver metastases, both AST and ALT ≤ 5× ULN Kidney: creatinine clearance (Ccr) ≥ 30mL/min in patients with multiple myeloma, Creatinine ≤ 1.5×ULN in other patients.

Coagulation:

International Normalized Ratio (INR) ≤ 1.5, Activated partial thromboplastin time (APTT) or prothrombin time (PT) ≤ 1.5× ULN.

corrected serum calcium ≤ 14 mg/dL (≤ 3.5 mmol/L). left ventricular ejection fraction (LVEF) ≥ 50%. 11. The patient and his/her spouse agree to take effective contraceptive measures (excluding contraception during the safe period) from the time of signing the informed consent form to 6 months after the last dose.

Exclusion Criteria:

1. Within 14 days before the first dose: received plasmapheresis; Treatment with > 10 mg of prednisone or equivalent doses of systemic corticosteroids per day for more than 3 consecutive days (short-term use for the prevention of contrast allergy can be enrolled).
2. Patients have received systemic anti-myeloma therapy or investigational drug therapy within 28 days or 5 half-lives (whichever is shorter) prior to the first dose; Radiotherapy within 14 days prior to the first dose.
3. Patients have received monoclonal antibody therapy within 30 days before the first dose.
4. Patients have received autologous hematopoietic stem cell transplantation within 100 days before the first dose.
5. Patients who have undergone allogeneic hematopoietic stem cell transplantation (HSCT) or have a history of solid organ transplantation.
6. Patients have received the same targeted therapy in the past (limited to phase Ia clinical trials).
7. Patient has symptomatic brain metastases or meningeal metastases.
8. The patient had symptomatic amyloidosis, active plasma cell leukemia, and active POEMS syndrome at the time of screening.
9. There is evidence of cardiovascular risk, including any of the following: a. QTcF interval ≥ 470 ms (QT interval must be corrected by Fridericia formula [QTcF]). b. Evidence of currently clinically significant, untreated arrhythmias, including clinically significant electrocardiogram abnormalities such as degree 2 (Mobitz type II) or degree 3 atrioventricular conduction (AV) block. c. History of myocardial infarction, acute coronary syndrome (including unstable angina pectoris), coronary angioplasty, or stenting or bypass grafting within 6 months prior to screening. d. Grade III or IV heart failure(New York Heart Association Functional Grading System). e. Uncontrolled severe hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥ 100 mmHg).
10. The patient has difficulty breathing or currently requires continuous oxygen therapy, or currently has active pneumonia or interstitial lung disease (except for mild cases as determined by the investigator).
11. The patient has a history of other primary malignancies, except the following: cured malignancies with a very low risk of recurrence within 5 years, such as skin basal cell carcinoma and skin squamous cell carcinoma, carcinoma in situ of the cervix or breast.
12. Patients have severe unhealed wound ulcers or fractures, or have undergone major surgery within 28 days prior to dosing or are expected to undergo surgery during the clinical study.
13. Previous history of allergy to any component or excipient of DXC006.
14. Active hepatitis B (HBV-DNA greater than the central upper limit of normal or HBV-DNA testing greater than 1000 copies /mL); Hepatitis C infection (positive for hepatitis C antigen or positive for hepatitis C RNA PCR).
15. Seropositive for human immunodeficiency virus (HIV); Active syphilis (patients with positive syphilis antibodies can be included); Possible active tuberculosis (chest imaging within 3 months prior to first dosing indicating active tuberculosis infection).
16. Patients had active bleeding within 30 days prior to screening, or were at risk of massive gastrointestinal bleeding or hemoptysis as determined by researchers; Or have inherited bleeding tendencies or coagulation disorders, or bleeding symptoms that require other medical intervention.
17. Severe arteriovenous thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism, occurred within 6 months before the first dose.
18. Female patients with a positive serological pregnancy test or who are breastfeeding.
19. Active infections requiring medical treatment (CTCAE≥2); Uncontrollable pleural fluid, ascites, pericardial effusion requiring repeated drainage;
20. Received live attenuated vaccine within 28 days before the first dose.
21. The patient has other conditions that the investigator or sponsor has determined may affect the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants that experienced dose limiting toxicities(DLTs) at given dose level. | 28 days
  Dose Limiting Toxicities (DLTs) In Order to Determine the Maximum Tolerated.
Number of participants with adverse events (AEs) | After first infusion of study drug, Through study completion an average of 1 year
  The adverse events will be evaluated in accordance with CTCAE v5.0. The investigator shall assess the relationship between the events and investigational product.

SECONDARY OUTCOMES:
Maximum observed serum or plasma concentration (Cmax) | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC006investigator shall assess the relationship between the events and investigational product.
Maximum serum drug time（Tmax） | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC006.
Apparent volume of distribution(Vd) | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC006.
Volume of distribution at steady state (Vss) | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC006.
Terminal phase elimination half life (t½) | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC006.
Area under the serum or plasma concentration time curve from 0 to the last measurable point (AUC0-t) | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC006.
Area under the serum or plasma concentration time curve from 0 to infinity (AUC0-inf) | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC006.
Clearance (CL) | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC006.
Anti-drug antibodies (ADA) | Through study completion an average of 1 year
  The titer,neutralizing activity and positive rate of anti-drug antibody (ADA).
Objective Response Rate (ORR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  As determined by the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, which will be complete response (CR) + partial response (PR).
Duration of response (DOR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  DOR is defined as the time from the date of the first documentation of response (confirmed CR or confirmed PR) to the date of the first documentation of PD or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) | om date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  PFS is defined as the time from the date of randomization to the earlier of the dates of the first documentation of progressive disease or death due to any cause.
Overall Survival (OS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  OS is defined as the time from the date of randomization to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Zhang Li, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT06224855/ICF_000.pdf